CLINICAL TRIAL: NCT06644079
Title: Window of Opportunity Pilot Study of Topical Tranexamic Acid for Cutaneous Squamous Cell Carcinoma
Brief Title: Window of Opportunity Study of Topical Tranexamic Acid for Cutaneous Squamous Cell Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study not moving forward due to upcoming PI departure
Sponsor: University of Florida (Other)
Collaborators: TXA Tech (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF-CUT-003
Record Dates: First submitted 2024-10-10; First posted 2024-10-16 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Cutaneous Squamous Cell Carcinoma
Keywords: topical tranexamic acid; cutaneous squamous cell carcinoma
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Topical tranexamic acid (Experimental)
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — Participants will self-apply topical tranexamic acid to the area where their disease is located 3 times daily for 21-28 days prior to their scheduled Moh's or excision surgery.

SUMMARY:
Tranexamic Acid (TXA) is a safe and effective antifibrinolytic drug used systemically to control bleeding and topically to treat melasma and rosacea. TXA suppresses the viability of multiple human/murine cancer cell lines and Plasmin formation, which prevents cleavage of the CDCP1 protein to a more oncogenic form. TXA appears to act through additional anticancer mechanisms that include reduction of S6K1 and STAT3 phosphorylation on sites required for their activation.

Uptake by cancer results in blockade of protein synthesis, and alter signaling through the amino acid-sensitive mTORC1/S6K1 and GCN2/eiF2a/ATF4 pathways. This is expected to induce autophagy, which may mediate some of the biological effects of TXA on cells. This effect of TXA is expected to be most prominent in cells that rely on high levels of basal protein synthesis such as cancer cells. Currently no clinical treatment in this space to spare or improve surgical outcomes.

Positive results could help reduce tumor size and suppress new cancer cell production before surgical interventions are taken. This treatment could improve the outcomes and treatments of people with skin cancer. If this window study is successful further studies will focus on patients with unresectable disease or those with lesions in areas difficult for surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age.
* A clinical diagnosis of squamous cell carcinoma confirmed pathologically through biopsy (shave, punch, or partial excision) consistent with Stage I or II cutaneous squamous cell carcinoma, including those but not limited to those with high-risk features by BWH staging criteria:

  1. Depth/invasion: > 2 mm thickness (Breslow thickness), Clark level ≥ IV, Perineural invasion
  2. Anatomic: Primary site ear
  3. Location: Primary site hair-bearing lip
  4. Differentiation: Poorly differentiated or undifferentiated
* Ability to apply topical treatment 3 times per day and record event times in a journal
* Use of other topical creams on affected areas
* Cutaneous squamous cell carcinoma secondary to immunosuppression and/or HIV allowed
* Subjects must not have more than one active malignancy at the time of enrollment (Subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen [as determined by the treating physician or approved by the PI] may be included).
* Written informed consent obtained from the subject and the subject agrees to comply with all the study-related procedures, such as ability to apply topical treatment 3 times per day and record times in a journal.
* Subjects of childbearing potential (SOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for at least 1 week after the last application of study treatment to minimize the risk of pregnancy. Prior to study enrollment, subjects of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy.

Exclusion Criteria:

* Allergy to TXA or any of its components
* Active skin infection at or near the tumor site
* Known stage III or IV disease
* Disease without measurable surface area following biopsy
* Subjects of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 1 week after the last application of study treatment.
* Subjects who are confirmed to be pregnant or breastfeeding.
* History of any other disease, metabolic dysfunction, clinical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for treatment complications, in the opinion of the treating physician.
* Prisoners or subjects who are involuntarily incarcerated, or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects who have a reduction in tumor size | 35 days
  Determine the percentage of subjects who have a reduction in tumor size at the time of definitive surgery, as compared to tumor size at baseline. This is measured by comparing the total tumor area before treatment with the total tumor area at the time of definitive surgery. Tumor area will be measured via images and will be calculated using length x width x height in mm.

SECONDARY OUTCOMES:
Difference in surgical defect size and tumor area at the time of surgery | At the time of surgery
  Determine the difference in surgical defect size and tumor area at the time of surgery
Maximal tumor reduction | 35 days
  Determine the maximal tumor volume by calculation of difference in total tumor volume between pre-treatment baseline and time of surgery. Tumor volume is calculated by direct visualization and measurements (in mm) of largest dimension in width x length x height of elevation off of skin surface.
Treatment compliance | 21-28 days
  Determine patient treatment compliance as measured by the percentage of doses applied out of total possible applications
Treatment tolerance | 21-28 days
  Determine patient treatment tolerance, as measured by patient reported description of irritation, difficulty in application, or other commentary on intolerance and by indirect evaluation of patient compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Bently Doonan, MD, MS, Principal Investigator — University of Florida